CLINICAL TRIAL: NCT00326729
Title: Fluid Shifts During Resuscitation: Impacts on Macrocirculation and Microcirculation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Montreal Burn Centre (Other)
Collaborators: Bristol-Myers Squibb (Industry); Canadian Anesthesiologists' Society (Other)
Other Study IDs: HD06-004
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-06-16 (Estimated); Status verified 2006-05

CONDITIONS: Burns
Keywords: burns; thermal injury; hemodynamics; microcirculation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Fluid resuscitation in burn patients is associated with major macrocirculatory and microcirculatory disturbances that have been poorly described. When done according to expert opinions, it is now rare to encounter the death of a patient due to an inadequate fluid resuscitation. Fluid resuscitation in burn patients is more opinion-based than evidence-based. Although burn admission to an intensive care facility is relatively rare, the burn patient is well suited to answer questions in the fluid resuscitation field because, as opposed to other critically ill patients:

1. investigators do have a time 'zero' for burn patients; they know exactly when the insult occurred;
2. apart from fluid resuscitation, the management of burn patients is uniform in the investigators' unit and is done according to various protocols;
3. the burn population is more uniform than the septic population making confounders and background noises less likely; and
4. as basic as it might sound, studying fluid resuscitation implies accomplishing a significant one; burn patients are the category of critically ill patients receiving the most important fluid resuscitation.

Studies that have addressed the question of fluid resuscitation in burn patients are quite numerous. However, they are either under-powered, dealing with various interventions or outcomes and sometimes of poor methodological quality.

Moving the investigators' focus from macrohemodynamic to microhemodynamic monitoring is now essential and due to recent technological advances, severe impairments in microcirculatory perfusion are now being recognized in various pathological states. What is now clear from various studies is the fact that even with restoring 'normal' macrocirculatory parameters, severe microcirculatory alterations can be seen.

This study is an integral part of a program aimed to explore different questions regarding fluid resuscitation in burn patients. The aim is to characterize changes in fluid shift, fluid accumulation, and vascular volumes after burn injury and also to study the effects of an artificial colloid on different macrocirculatory and microcirculatory parameters. The primary end points are:

1. fluid accumulation during the initial phase; and
2. short term effects of colloids on macrocirculatory and microcirculatory parameters.

This study will collect data on macro- and microcirculation derived from current monitoring systems. Data (see below) will be collected at defined time points and before and after the first two fluid challenges. If the fluid challenge occurs in a one hour time frame of a defined time point, only one assessment will be done.

1. At defined time points: a set of data (see below) will be collected by the research team at baseline, 6, 12, 18, 24, 36, 48 and 72 hours after burn injury. Baseline values will be the ones obtained immediately after consent.
2. Fluid challenges: Burn patients often require additional fluid bolus to maintain hemodynamic stability because of the following reasons: hypotension; decreased urine output (less than 0.5 ml/kg/hour); uncorrected metabolic acidosis; rhabdomyolysis; increasing hematocrit; or any other clinical reason according to the attending physician.

In this study, the two first fluid challenges will be allocated according to a random list. One bolus will be Pentaspan (500 ml) and the other will be a crystalloid solution (Ringer's lactate 1000 ml). These two alternatives represent a true equipoise as they are equally acceptable because choosing one of them depends on the preference of the attending physician. Fluid challenges will be allocated using a randomised short block cross-over sequence.

The following parameters will be measured at a fixed time and before and after the fluid challenges using different techniques.

Parameters:

Intrathoracic blood volume, extravascular lung water, total blood volume; extracellular edema; intraventricular preload, ventricular volumes, diastolic function; cardiac output; mixed venous saturation; oncotic pressure; microcirculatory assessment: number and diameter of capillaries, proportion of perfusion, and flow velocities.

This is an observational, one-group study aimed at describing macrocirculation and microcirculation parameters in a burn patient population. The investigators arbitrarily plan to enroll 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Major thermal, electrical, or chemical burns
* Admission to the burn unit within 6 hours after burn
* Burned surface area over 20% or equivalent
* Signed consent by the patient or relative
* Commitment to full maximal support

Exclusion Criteria:

* Patient under 18 years old
* Patient over 80 years old
* Pregnancy
* Chronic renal failure requiring dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: David Bracco, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal; Marc-Jacques Dubois, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal
Locations (1):
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada